CLINICAL TRIAL: NCT06635590
Title: The Impact of Hyperkalemia-Induced ECG and ECHO Findings on Early and Late Mortality in Patients With Chronic Kidney Disease
Brief Title: Chronic Kidney Disease, Hyperkalemia and Echocardiographic Changes
Status: Recruiting | Type: Observational
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Sponsor
Other Study IDs: CKD ,HYPERKALEMIA AND ECHO
Record Dates: First submitted 2024-10-08; First posted 2024-10-10 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: Chronic Kidney Disease (CKD); Hyperkalemia; Hemodialysis
Keywords: echocardiography; ECG; chronic kidney disease; hyperkalemia
MeSH Terms: conditions — Renal Insufficiency, Chronic; Hyperkalemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hyperkalemia: Study is planned as only 1 group of patient with hyperkalemia. Pre and post treatment data obtained from patients via ECG, ECHO and laboratory values will be recorded and evaluated in terms of literature. Patient-based findings will also be recorded and evaluated.

SUMMARY:
Patients with CKD ( eGFR < <60 mL/min/1,73 m2) presenting to emergency department with isolated hyperkalemia will be study population. Pre and post treatment ECG and echocardiographic findings will be recorded. Investigator will not intervene with the treatment decision of responsible physician and will not delay any intervetion or treatment for the sake of study.

Data will be compared in terms of ECHO and ECG findings depending on hyperkalemia level and response to treatment.

DETAILED DESCRIPTION:
In this study, the ECG and echocardiography (ECHO) findings in patients with chronic kidney failure who present to the Etlik City Hospital Emergency Medicine Department will be recorded and compared with literature. Echocardiography is a rapid, reliable, and non-invasive examination widely used by physicians for the monitoring of critically ill patients in emergency departments and intensive care units worldwide.

For patients with known chronic kidney failure brought to the emergency department, a blood sample (blood gas and/or biochemistry) will be taken for potassium measurement. Subsequently, an ECG, which is a quick and non-invasive test, will be performed, followed by an ECHO, also a quick and non-invasive test, conducted by an experienced physician. The physician performing the ECHO will not be involved in the treatment process. ECG and ECHO findings will be recorded and compared before and after treatment. Patient mortality will be monitored at 24 hours, 7 days, and 30 days, and other causes of mortality will be excluded. The relationship between ECG and ECHO findings and mortality will be statistically investigated.

Based on the premise that hyperkalemia can cause cardiac arrest during diastole, it is hypothesized that there may be right ventricular enlargement in patients with ECG findings indicative of hyperkalemia. In animal studies, echocardiography results during resuscitation have shown right ventricular enlargement in animals with hyperkalemia. Based on this information, we believe that echocardiography findings in hyperkalemic patients may be associated with mortality, and that the combined use of echocardiography and ECG may be effective in predicting mortality

ELIGIBILITY:
Inclusion Criteria:

1. Patients over 18 years old
2. Chronic kidney disease patients with eGFR < 60 mL/min/1.73 m²
3. Patients with hyperkalemia detected in the emergency department
4. Patients willing to participate in the study and who sign the consent form

Exclusion Criteria:

1. Patients under 18 years old
2. Patients who do not wish to participate in the study
3. Patients without chronic kidney damage
4. Patients without detected hyperkalemia
5. Patients needing cardiopulmonary resuscitation due to hyperkalemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with chronic kidney disease presenting to emergency department and having isolated hyperkalemia with or without ECG changes
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
ECHO changes | from enrollment to the end of follow up duration of 30 days
  Describing echocardiograhic (ECHO) changes of isolated hyperkalemia in patients with chronic kidney disease (CKD)

CONTACTS AND LOCATIONS:
Overall Officials: gulsen akcay, ass. prof., Study Director — ass. prof. of organization
Locations (1):
- Etlik City Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Weiss JN, Qu Z, Shivkumar K. Electrophysiology of Hypokalemia and Hyperkalemia. Circ Arrhythm Electrophysiol. 2017 Mar;10(3):e004667. doi: 10.1161/CIRCEP.116.004667. No abstract available. PMID 28314851
- [Result] Kim MJ, Valerio C, Knobloch GK. Potassium Disorders: Hypokalemia and Hyperkalemia. Am Fam Physician. 2023 Jan;107(1):59-70. PMID 36689973
- [Result] Piner A, Spangler R. Disorders of Potassium. Emerg Med Clin North Am. 2023 Nov;41(4):711-728. doi: 10.1016/j.emc.2023.07.005. PMID 37758419